CLINICAL TRIAL: NCT04023435
Title: Pain Neuroscience Education for Depression
Acronym: PNEdepress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Ambrose University (Other)
Responsible Party: Principal Investigator, Kevin Farrell, Professor and Chair, Orthopaedic Residency Program in Physical Therapy, St. Ambrose University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1819307
Record Dates: First submitted 2019-07-11; First posted 2019-07-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Chronic Low-back Pain; Depression
Keywords: chronic; Low-Back Pain; Depression
MeSH Terms: conditions — Depression; Bronchiolitis Obliterans Syndrome; Low Back Pain

STUDY DESIGN:
Intervention Model Description: This will be a pre- and post-intervention convenience sample of consecutive patients with chronic LBP (pain > 6 months) meeting the inclusion criteria, attending outpatient PT. On initial examination, intake data and information will be collected prior to PNE and immediately following PNE.
Masking Description: No other parties will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PNE education (Experimental): All subjects will be tested before and after receiving PNE education
  Interventions: Other: PNE edcuation

INTERVENTIONS:
Other: PNE edcuation — The PNE session will last 30 minutes and will be delivered in a one-on-one educational format with a clinician using prepared images, drawings and metaphors. The 30-minute PNE session was chosen to reflect a clinically meaningful intervention in a typical allocated time frame in clinical practice. The content of the PNE is described in detail elsewhere, using a metaphors to explain various aspects of pain including sensitization of the peripheral and central nervous system (sensitive alarm system metaphor); spreading pain (nosy neighbors metaphor); increases problems with focus and concentration (brain meeting metaphor) and difficulty with fatigue and sleep (lion metaphor).

SUMMARY:
This study will look at the effects of Pain Neuroscience Education on a Depression outcome tool in patients with chronic low back pain.

DETAILED DESCRIPTION:
Pain and depression have been shown to be interrelated, especially chronic pain: people in chronic pain develop depression and people with depression develop chronic pain. In light of this coexistence it is not surprising that current best-evidence for depression and chronic pain shows significant overlap which includes primarily some type of cognitive intervention, aerobic exercise, and skilled delivery of medication including selective-serotonin-reuptake-inhibitors and/or membrane stabilizers. Current best-evidence regarding musculoskeletal pain provides strong support for Pain Neuroscience Education (PNE) to positively influence pain ratings, dysfunction, and limitations in movement, pain knowledge and healthcare utilization. Additionally, PNE has shown to powerfully influence psychosocial issues that powerfully influence pain and depression: fear-avoidance and pain catastrophization. Evidence is lacking in whether PNE could also influence depression ratings. The purpose of this study is to examine the immediate effect of PNE on pain, function, and depressive symptoms (using the Patient Health Questionnaire - PHQ-9) in patients attending PT for chronic low back pain (LBP).

This will be a pre- and post-intervention convenience sample of consecutive patients with chronic LBP (pain > 6 months) meeting the inclusion criteria, attending outpatient PT. On initial examination, intake data and information will be collected prior to PNE and immediately following PNE.

ELIGIBILITY:
Inclusion Criteria:

* adults over the age of 18
* presenting at PT with a primary complaint of LBP
* LBP being present for 6 months or more
* fluent in English
* willing to participate in the study.

Exclusion Criteria:

* are under age 18 (minor)
* had undergone lumbar surgery
* cannot read or understand the English language
* presents with any cognitive deficits rendering them unsuitable for PNE (i.e., stroke, traumatic brain injury, etc.)
* decline to participate
* present with a medical etiology (red flag) associated with their LBP.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Low back pain rating | within a single, 90 minute session
  Numeric Pain Rating Scale for Back Pain (0 = no pain and 10 = worst pain). The minimal detectable change (MDC) for the NPRS for low back pain is reported to be 2.0.
Pain Catastrophization Scale | within a single, 90 minute session
  The PCS is a self-report questionnaire assessing inappropriate coping strategies and catastrophic thinking about pain and injury. on a 13-item, 5-point Likert scale with higher scores indicating elevated levels of catastrophizing.
revised Pain Neurophysiology Questionnaire - rNPQ | within a single, 90 minute session
  The NPQ measures the neurophysiology knowledge of patients and healthcare personnel. The original NPQ is a 19-item questionnaire requesting 'true'; 'false'; or 'not sure' answers to statements, with higher scores indicating more correct answers.
Patient Health Questionnaire - PHQ-9 | within a single, 90 minute session
  The PHQ-9 is the nine item depression scale

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Farrell, Principal Investigator — St. Ambrose University
Locations (1):
- Kevin Farrell, Davenport, Iowa, United States

IPD SHARING:
Plan to Share IPD: No